CLINICAL TRIAL: NCT05779410
Title: Effects of Vitamin D Supplementation on Biochemical Responses and Aerobic Capacity After Strenuous Endurance Exercise
Brief Title: Vitamin D in Healthy Adults After Strenuous Endurance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Panion & BF Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202010026; A-107-077 (Other Grant/Funding Number: Panion & BF Biotech Inc.)
Record Dates: First submitted 2023-02-20; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Healthy male participants were divided into vitamin D group and placebo group.
Who Masked: Participant, Investigator
Masking Description: A double-blind, matched-pair study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental)
  Interventions: Dietary Supplement: Vitamin D
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Medium-chain triglycerides

INTERVENTIONS:
Dietary Supplement: Vitamin D — Participants received 5,000 IU of vitamin D orally twice daily for 4 weeks
  Other Names: Liquid Shield Vitamin D3+E
  Arms: Vitamin D group
Dietary Supplement: Medium-chain triglycerides — Participants received the same amount of placebo matching vitamin D orally twice daily for 4 weeks
  Arms: Placebo group

SUMMARY:
The purpose of this study was to investigate the effects of vitamin D supplementation on biochemical response and aerobic capacity after strenuous endurance exercise (SEE).

DETAILED DESCRIPTION:
All participants conducted a graded exercise test on an ergometric bicycle to determine the maximal oxygen consumption (VO2max) before and after supplementation, and the speed equivalent to 65% VO2max was conducted for a SEE test by ergometric bicycle for 2 hours, followed by increasing 100 RPM until exhaustion. Venous blood samples were drawn before, immediately after, 2-hour after, 4-hour after, 8-hour after, and 24-hour after the SEE test to determine the concentrations of biomarkers. Data was analyzed by Two-way mixed design ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* The volunteers included have conditions as stated below :

  1. no history of cardiovascular, liver, kidney and diabetes disease
  2. no acute sport injury
  3. male adult whose concentration of 25(OH)D is under 30 ng/mL, and maximal oxygen consumption is over 40 ml/kg/min
  4. did not participated in any clinical trials or research in the last 3 months before our experiment
  5. no supplements were taken during the experimental period
  6. were requested to maintain their regular daily life style and avoid alcohol intake

Exclusion Criteria:

* The volunteers were excluded if they have the situation stated below:

  1. history of cardiovascular, liver, kidney and diabetes disease
  2. acute sport injury
  3. their concentration of 25(OH)D is over 30 ng/mL, or maximal oxygen consumption is under 40 ml/kg/min
  4. participated in any clinical trials or experimental research in the last 3 months before our experiment
  5. taking supplement during the experimental period
  6. did not maintain their regular eating habit or drink alcohol

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The sample size is small due to the limited research funding. Additionally, considering the sports ability between men and women is significantly different, there would be a large standard deviation if we include both males and females. Thus our study includes male subjects only.
Enrollment: 35 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Concentration of Neutrophil | before exercise
Concentration ofNeutrophil | immediately after exercise
Concentration of Neutrophil | 2-hour after exercise
Concentration of Neutrophil | 4-hour after exercise
Concentration of Neutrophil | 8-hour after exercise
Concentration of Neutrophil | 24-hour after exercise
Concentration of eosinophil | before exercise
Concentration of eosinophil | immediately after exercise
Concentration of eosinophil | 2-hour after exercise
Concentration of eosinophil | 4-hour after exercise
Concentration of eosinophil | 8-hour after exercise
Concentration of eosinophil | 24-hour after exercise
Concentration of basophil | before exercise
Concentration of basophil | immediately after exercise
Concentration of basophil | 2-hour after exercise
Concentration of basophil | 4-hour after exercise
Concentration of basophil | 8-hour after exercise
Concentration of basophil | 24-hour after exercise
Concentration of monocyte | before exercise
Concentration of monocyte | immediately after exercise
Concentration of monocyte | 2-hour after exercise
Concentration of monocyte | 4-hour after exercise
Concentration of monocyte | 8-hour after exercise
Concentration of monocyte | 24-hour after exercise
Concentration of lymphocyte | before exercise
Concentration of lymphocyte | immediately after exercise
Concentration of lymphocyte | 2-hour after exercise
Concentration of lymphocyte | 4-hour after exercise
Concentration of lymphocyte | 8-hour after exercise
Concentration of lymphocyte | 24-hour after exercise
Concentration of CD4+ | before exercise
Concentration of CD4+ | immediately after exercise
Concentration of CD4+ | 2-hour after exercise
Concentration of CD4+ | 4-hour after exercise
Concentration of CD4+ | 8-hour after exercise
Concentration of CD4+ | 24-hour after exercise
Concentration of CD8+ | before exercise
Concentration of CD8+ | immediately after exercise
Concentration of CD8+ | 2-hour after exercise
Concentration of CD8+ | 4-hour after exercise
Concentration of CD8+ | 8-hour after exercise
Concentration of CD8+ | 24-hour after exercise
Concentration of CD19+ | before exercise
Concentration of CD19+ | immediately after exercise
Concentration of CD19+ | 2-hour after exercise
Concentration of CD19+ | 4-hour after exercise
Concentration of CD19+ | 8-hour after exercise
Concentration of CD19+ | 24-hour after exercise
Concentration of CD56+ | before exercise
Concentration of CD56+ | immediately after exercise
Concentration of CD56+ | 2-hour after exercise
Concentration of CD56+ | 4-hour after exercise
Concentration of CD56+ | 8-hour after exercise
Concentration of CD56+ | 24-hour after exercise
Concentration of IgA | before exercise
Concentration of IgA | immediately after exercise
Concentration of IgA | 2-hour after exercise
Concentration of IgA | 4-hour after exercise
Concentration of IgA | 8-hour after exercise
Concentration of IgA | 24-hour after exercise
Concentration of Cathelicidin | before exercise
Concentration of Cathelicidin | immediately after exercise
Concentration of Cathelicidin | 2-hour after exercise
Concentration of Cathelicidin | 4-hour after exercise
Concentration of Cathelicidin | 8-hour after exercise
Concentration of Cathelicidin | 24-hour after exercise
Concentration of TNF-α | before exercise
Concentration of TNF-α | immediately after exercise
Concentration of TNF-α | 2-hour after exercise
Concentration of TNF-α | 4-hour after exercise
Concentration of TNF-α | 8-hour after exercise
Concentration of TNF-α | 24-hour after exercise
Concentration of IL-1β | before exercise
Concentration of IL-1β | immediately after exercise
Concentration of IL-1β | 2-hour after exercise
Concentration of IL-1β | 4-hour after exercise
Concentration of IL-1β | 8-hour after exercise
Concentration of IL-1β | 24-hour after exercise
Concentration of IFN-γ | before exercise
Concentration of IFN-γ | immediately after exercise
Concentration of IFN-γ | 2-hour after exercise
Concentration of IFN-γ | 4-hour after exercise
Concentration of IFN-γ | 8-hour after exercise
Concentration of IFN-γ | 24-hour after exercise
Concentration of IL-2 | before exercise
Concentration of IL-2 | immediately after exercise
Concentration of IL-2 | 2-hour after exercise
Concentration of IL-2 | 4-hour after exercise
Concentration of IL-2 | 8-hour after exercise
Concentration of IL-2 | 24-hour after exercise
Concentration of IL-4 | before exercise
Concentration of IL-4 | immediately after exercise
Concentration of IL-4 | 2-hour after exercise
Concentration of IL-4 | 4-hour after exercise
Concentration of IL-4 | 8-hour after exercise
Concentration of IL-4 | 24-hour after exercise
Concentration of IL-8 | before exercise
Concentration of IL-8 | immediately after exercise
Concentration of IL-8 | 2-hour after exercise
Concentration of IL-8 | 4-hour after exercise
Concentration of IL-8 | 8-hour after exercise
Concentration of IL-8 | 24-hour after exercise
Concentration of IL-10 | before exercise
Concentration of IL-10 | immediately after exercise
Concentration of IL-10 | 2-hour after exercise
Concentration of IL-10 | 4-hour after exercise
Concentration of IL-10 | 8-hour after exercise
Concentration of IL-10 | 24-hour after exercise
Concentration of TBARS | before exercise
Concentration of TBARS | immediately after exercise
Concentration of TBARS | 2-hour after exercise
Concentration of TBARS | 4-hour after exercise
Concentration of TBARS | 8-hour after exercise
Concentration of TBARS | 24-hour after exercise
Concentration of PC | before exercise
Concentration of PC | immediately after exercise
Concentration of PC | 2-hour after exercise
Concentration of PC | 4-hour after exercise
Concentration of PC | 8-hour after exercise
Concentration of PC | 24-hour after exercise
Concentration of SOD | before exercise
Concentration of SOD | immediately after exercise
Concentration of SOD | 2-hour after exercise
Concentration of SOD | 4-hour after exercise
Concentration of SOD | 8-hour after exercise
Concentration of SOD | 24-hour after exercise
Concentration of catalase | before exercise
Concentration of catalase | immediately after exercise
Concentration of catalase | 2-hour after exercise
Concentration of catalase | 4-hour after exercise
Concentration of catalase | 8-hour after exercise
Concentration of catalase | 24-hour after exercise
Concentration of GPx | before exercise
Concentration of GPx | immediately after exercise
Concentration of GPx | 2-hour after exercise
Concentration of GPx | 4-hour after exercise
Concentration of GPx | 8-hour after exercise
Concentration of GPx | 24-hour after exercise
Concentration of CK | before exercise
Concentration of CK | immediately after exercise
Concentration of CK | 2-hour after exercise
Concentration of CK | 4-hour after exercise
Concentration of CK | 8-hour after exercise
Concentration of CK | 24-hour after exercise
Concentration of LDH | before exercise
Concentration of LDH | immediately after exercise
Concentration of LDH | 2-hour after exercise
Concentration of LDH | 4-hour after exercise
Concentration of LDH | 8-hour after exercise
Concentration of LDH | 24-hour after exercise
Concentration of IL-6 | before exercise
Concentration of IL-6 | immediately after exercise
Concentration of IL-6 | 2-hour after exercise
Concentration of IL-6 | 4-hour after exercise
Concentration of IL-6 | 8-hour after exercise
Concentration of IL-6 | 24-hour after exercise
Concentration of CRP | before exercise
Concentration of CRP | immediately after exercise
Concentration of CRP | 2-hour after exercise
Concentration of CRP | 4-hour after exercise
Concentration of CRP | 8-hour after exercise
Concentration of CRP | 24-hour after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan